CLINICAL TRIAL: NCT02644304
Title: Clomiphene Citrate Plus Cabergoline Versus Clomiphene Citrate Alone in Treatment of Polycystic Ovary Syndrome Associated Infertility
Brief Title: Clomiphene Citrate Plus Cabergoline in Treatment of Polycystic Ovary Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Kamal Mohamed Zahran, Dr, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CC in PCOS
Record Dates: First submitted 2015-10-13; First posted 2015-12-31 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Female Reproductive Problem
MeSH Terms: interventions — Clomiphene; Cabergoline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clomiphene citrate plus cabergoline (Active Comparator): This group will receive Clomiphene citrate 50 mg tablet twice daily from the second day of menses to the sixth day plus cabergoline 0.25 mg from second day every 3 days (4 doses only)
  Interventions: Drug: Clomiphene citrate; Drug: Cabergoline
- Clomiphene citrate plus placebo (Active Comparator): This group will receive Clomiphene citrate 50 mg tablet twice daily from the second day of menses to the sixth day plus placebo tablets from second day every 3 days (4 doses only)
  Interventions: Drug: Clomiphene citrate; Other: Placebo

INTERVENTIONS:
Drug: Clomiphene citrate — 50 mg tablet twice daily from the second day of menses to the sixth day
Drug: Cabergoline — Cabergoline 0.25 mg (half tablet) every 3 days (4 doses).
  Arms: Clomiphene citrate plus cabergoline
Other: Placebo — placebo(half tablet) every 3 days (4 doses).
  Arms: Clomiphene citrate plus placebo

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common endocrine disorder of reproductive aged women and affects approximately 5-12 % of the female population.

In 2003 in Rotterdam , Rotterdam diagnostic criteria were redefined PCOS as affected individuals must have two out of the following three criteria:

1. Oligo- and/or anovulation, (ovulation occurs less than once every 35 days).
2. Hyperandrogenism, clinical signs include hirsutism, acne, alopecia, and frank virilization, while chemical indicators include raised concentrations of total testosterone and androstenedione , and elevated free androgen index.
3. Polycystic ovaries on sonographic examination, presence of 12 or more follicles in either ovary measuring 2-9 mm in diameter, increased ovarian volume more than 10 cm3 and/or increase in stromal echogenicity. Clearly, according to the Rotterdam diagnostic criteria, the majority of women with PCOS can be diagnosed without the need of laboratory examinations.

Clomiphene citrate (CC) is still the first-line medication for the induction of ovulation. It is an anti-estrogenic compound made up of two isomers, enclomiphene and zuclomiphene; the latter being the more potent of the two. It is a non-steroidal compound closely resembling estrogen. CC acts by blocking estrogen receptors, particularly in the hypothalamus, thereby signaling a lack of circulating estrogens and inducing a change in the pulsatile release of gonadotrophin-releasing hormone (GnRH). This induces release of follicle stimulating hormone from the anterior pituitary and is often enough to set the cycle of events leading to ovulation into motion.

Cabergoline, ergot-derived dopamine agonists with a very long half life, is an effective prolactin suppressor. Cabergoline oral administration contains a weekly dose of 0.5 - 3 mg, which could be increased, if needed, to twice a week. This medicine has slight dopamine agonistic side effects, headache being the most common one. Treatment in the very beginning should start with a partial dose (half a pill) at bedtime with a small amount of food. Low incidence of side effects and its weekly dose has made Cabergoline a choice drug for treatment of related diseases.

ELIGIBILITY:
Inclusion Criteria:

* 2 or more of PCOS signs according to Rotterdam diagnostic criteria (2003).-
* Primary or secondary infertility.-
* Absence of galactorrhoea
* Normal serum prolactin or slightly elevated (up to 50 ng/dl)
* Normal hysterosalpingography
* Normal spermogram

Exclusion Criteria:

* Women on other line of treatment as aromatase inhibitors, gonadotrophins, or tamoxifen.
* Known hypersensitivity for Clomiphene citrate or cabergoline.
* Other factors of infertility as tubal factor, uterine factor or male factor.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Size of mature follicles (mm). | 1 year

SECONDARY OUTCOMES:
Number of pregnancy | 1 year
Number of mature follicles (mm) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt